CLINICAL TRIAL: NCT04158726
Title: Integrating Geriatric Assessment for Older Patients Diagnosed With Acute Myelogenous Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 422 AML GA
Record Dates: First submitted 2019-11-01; First posted 2019-11-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: modified Geriatric Assessment (mGA) — The mGA, administered via patient self-report on a touchscreen computer, as well as the real-time use and utility by clinicians and the correlation of mGA results on treatment decision-making.

SUMMARY:
Despite the suggestions that GA and frailty indices could be used to guide therapy selection, the ability to effectively incorporate the use of GA in older patients diagnosed with AML in a real-world clinic environment has not yet been established. Thus, in this study, the investigators seek to describe the feasibility of using this shorter GA tool, the mGA, administered via patient self-report on a touchscreen computer, as well as the real-time use and utility by clinicians and the correlation of mGA results on treatment decision-making.

DETAILED DESCRIPTION:
This outcomes study has a two-part intervention that includes 1) provider education and 2) patient and provider use of Carevive Treatment Care Planning technology. The provider education component of the intervention highlights evidenced guidelines and investigational agents in the treatment of AML in older adults. The Carevive CPS will be used for the second component of the intervention. The results of this study will provide important information about drivers of treatment decision-making and practice patterns, feasibility of a technology platform to incorporate important, but under-utilized components of value-based care into practice, and healthcare utilization data.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be adults ages 18 years of age or older.
* Patient participants must have a diagnosis of AML.
* Patients may be newly diagnosed, needing a new line of therapy and have not yet made a treatment decision, or on treatment and being assessed for potential new treatment
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The correlation of mGA for patients with AML on clinical outcomes at three months post treatment decision making. | 3 months
  Clinical outcomes include time on treatment, adherence to the prescribed treatment, quality of life (QoL), and patient side effects. Providers will review results of the mGA at a treatment decision visit and indicate if the mGA results influenced the treatment selection. Chart abstraction will be conducted at a 3-month post treatment planning visit time point to confirm treatment given. Baseline and 3-month QoL and symptom assessment measures will be collected and change over time will be analyzed. Comparisons of change in QoL and symptoms over 3 months, total time on treatment, and adherence among fit, intermediate, and frail groups will be made.

SECONDARY OUTCOMES:
Review of Real-world clinician practice patterns of hematologists managing older patients with AML (age>60), | 3 months
  Quantitative measures include data collected by the Carevive CPS platform to describe treatment practice patterns of hematologists caring for older patients with AML at three study sites. At baseline, and then again as part of participating clinicians' exit interview, each clinician will complete a survey that asks about his/her behaviors related to assessment and management of their older AML patients.

OTHER OUTCOMES:
Satisfaction (usability, acceptability, feasibility and utility) of incorporating electronic mGA into routine clinical care will be evaluated at baseline and each clinic visit.A comprehensive survey will be utilized to capture these outcomes. | 3 months
  Usability and acceptability of the electronic mGA is measured by both patients and providers using surveys after the visit. Feasibility of the mGA is assessed at the patient level and focuses on the patient's ability to complete the assessment via an electronic tablet prior to their visit without assistance. These measures will be collected using one comprehensive survey
Change in the hematologists' knowledge, skills and attitudes from baseline following continuing education modules viewed by providers. | 3 months
  Clinicians will complete a pre-test and a post-test questionnaire, allowing for the determination of clinician competency to optimally manage older patients with AML based on GA screening. The comparisons will assess changes in knowledge, skills and attitudes as a direct result of the training. Surveys will be completed capturing the results and will be compared at the different timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Wujcik, PhD,RN, Principal Investigator — Carevive Systems, Inc.
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No